CLINICAL TRIAL: NCT03718078
Title: Essai Clinique Pour Une Endomicroscopie Robotisée Dans la redéfinition Des Stratégies d'ExérèsE (PERSÉE) appliquée à la Chirurgie Hépatique
Brief Title: Robotic Endomicroscopy to Better Define Resection Strategies Applied to Hepatic Surgery
Acronym: PERSEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MKT-2018-PERSEE-02-DIG; 2018-A02619-46 (Other: ID-RCB)
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Hepatocarcinoma; Hepatic Metastasis; Hepatic Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Confocal Laser Endomicroscopy (Experimental): lt includes patients will undergo probe-based Confocal Laser Endomicroscopy during laparoscopic hepatic masses resection.
  Interventions: Device: Confocal Laser Endomicroscopy

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy — The study is divided in two parts. For the two parts, patients will receive an intravenous injection of indocyanine green:
  1. Ex vivo study
     - Images/sequences of normal and abnormal hepatic tissues and surgical margins will be acquired on surgical specimens
  2. In vivo study - Intra-operative pCLE imaging will be performed on hepatic masses and surgical margins
  Other Names: probe-based Confocal Laser Endomicroscopy; CelioFlex UHD 5 probe; Viziobot-P; GastroFlex UHD probe; Cellvizio 100 series; pCLE; Confocal Miniprobes

SUMMARY:
This study aims at assessing the feasibility of Probe-based Confocal Laser Endomicroscopy (pCLE) during laparoscopic hepatic masses resection for intra-operative characterisation of hepatic masses and surgical margins assessment.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer and third leading cause of cancer deaths in the Western countries. In France, 45.000 new patients develop colorectal cancer every year. The liver is the most common organ targeted by CRLM, representing 50%. Approximately, 15-25% of colorectal cancer patients have synchronous CRLM at initial workup, and 20-30% patients sustain subsequent liver metastases within few years following diagnosis.

The strategy for colorectal cancer liver metastasis resection and liver cancer has evolved to a parenchymatic sparing procedure. This technic aims to minimize surgical margins width while removing the tumor. Therefore, the current standard for resection margins is a margin width superior to 1mm. However, there is still a debate concerning the margin width. Indeed, with modern chemotherapy, several studies reported no statistical differences in the overall survival between R0 patients and R1 patients treated with chemotherapy. However, in order to preserve patients from chemotherapy treatments' adverse effects an intra-operative microscopic assessment of surgical margins should be set up in order to reduce R1 margins occurrence.

Ex vivo study:

Surgical specimens obtained during hepatectomy will be imaged to generate an atlas of pCLE images.

In vivo study:

Intraoperative characterization of sub-capsular hepatic masses and surgical margins will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Scheduled for a surgical resection of hepatic masses
* Provided signed informed consent

Exclusion Criteria:

* Allergy to Indocyanine green (ICG)
* Kidney failure
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-01-07 (Estimated); Study Completion 2020-01-07 (Estimated)

PRIMARY OUTCOMES:
malignant pCLE criteria | 1 year
  Definition of pCLE criteria for normal and malignant hepatic tissues

SECONDARY OUTCOMES:
pathological pCLE criteria | 1 year
  Definition of pCLE criteria for pathological hepatic parenchyma (non tumoral)
Ease of use of the endomicroscopy device | 1 year
  The ease of use of the endomicroscopy device will be assessed using a questionnaire that the surgeon will fill at the end of each procedure
Audio/video telecommunication quality | 1 year
  The telecommunication quality will be assessed using a questionnaire that the surgeon and the anatomopathologist will fill at the end of each procedure
Number of participants with CLE imaging-related adverse events as assessed by CTCAE v5.0 | 1 year
  The device safety will be measured by assessing the occurence and severity of adverse events during the study
Stability and reproducibility of images/sequences during procedures | 1 year
  The stability and reproducibility of endomicroscopy images will be assessed using a questionnaire that the surgeon and the anatomopathologist will fill at the end of each procedure
pCLE criteria diagnostic performance | 1 year
  The diagnostic performance of identified pCLE criteria will be expressed by their sensitivities, specificities, negative predictive value and positive predictive value.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Mutualiste Montsouris, Paris, France